CLINICAL TRIAL: NCT06625359
Title: Efficacy of High-dose Chemotherapy with Thiotepa, Busulfan, and Cyclophosphamide Before Autologous Stem Cell Transplantation in Patients with Primary/secondary Central Nervous System Lymphoma
Brief Title: High-dose Chemotherapy with Thiotepa, Busulfan, and Cyclophosphamide Followed by Autologous Stem Cell Transplantation in Central Nervous System Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, YOUNGIL KOH, Professor doctor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-1503-129-659
Record Dates: First submitted 2024-09-30; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Central Nervous System Lymphoma
Keywords: PCNSL; SCNSL; high-dose chemotherapy followed by autoSCT; Thiotepa, Busulfan, Cyclophosphamide
MeSH Terms: interventions — Thiotepa; Tubercidin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Patients with histologically confirmed primary central nervous system lymphoma or secondary CNS lymphoma defined as either synchronous CNS involvement of sys- temic NHL or as a site of recurrence in a patient s with a history of systemic NHL
  * Patients who achieved remission after first line chemotherapy and/or WBRT, or who experience relapse of PCNSL/SCNLS.
  * Patients who have not previously received therapy with high high-dose chemotherapy and stem cell transplantatitransplantation.
  * The performance st atus of the patients should be 2 or less by ECOG performance scale.
  * Patients should not have major illness or organ failure incompatible with autologous stem cell transplantation.
  Interventions: Drug: Thiotepa in conditioning before transplantation

INTERVENTIONS:
Drug: Thiotepa in conditioning before transplantation — For patients with ECOG PS 0 or 1 For patients with ECOG PS 0 or 1 and age < 60 years old, conditioning regimen before autologous stem cell transplantation consists of thiotepa, bulsulfan, and cyclophosphamide from day -9. Beginning on day -9 and through day -7, each patient was treated with thiotepa (200mg/m m2 IV per day). On days -6 to -4, patients received bulsulfan (2.7mg/kg IV over 3 hours per day every). Bulsulfan-related seizure prophylaxis was given with levetriacetam (1500mg loading on day -6, 500mg twice daily on days -5 to -3). On days -3 and -2, cyclophosphamide (60mg/kg IV per day) was given given.
  Patients with ECOG PS 2 or age ≥ 60 years old received bulsulfan (3.2mg/kg IV over 3 hours per day for 2 days) resulting in 8 days regimen.
  Other Names: high-dose CTx with TBC, followed by auto-SCT

SUMMARY:
The involvement of the central nervous system (CNS) by non-Hodgkin lymphoma (NHL) has carried a poor prognosis. For both of primary central nervous system lymphoma (PCNSL) and secondary central nervous system lymphoma (SCNSL), high-dose methotrexate (HD- MTX) based chemotherapy and combined modality have significantly improved the previously poor response rates and prognosis. However, in PCNSL, relapse rates have remained high, with only 20% to 30% patients achieving a durable long-term remission after HD-MTX. The combination with whole-brain radiotherapy (WBRT) has resulted in higher disease-free and overall survival rates, but it has also been associated with severe neurotoxicity. Patients with SCNSL fare the worst, typically succumbing to disease within median 2.5 to 4 months with 1-year survival rates of only 25%.

Because of these dismal outcomes, intensification of the high-dose chemotherapy (HDC)with autologous stem cell transplantation (autoSCT) has been explored for PCNSL and SCNSL as salvage treatment in patients with refractory or relapsed disease, and as consolidation after primary chemotherapy, replacing or preceding WBRT. Thiotepa, busulfan, and cyclophosphamide (TBC) have significant penetration of blood-brain barrier as shown in several pharmacokinetic studies. Thus, combination of these 3 agents was proposed as one high-dose chemotherapy regimen to achieve therapeutic concentrations in the lymphoma tissue in chemotherapy sanctuaries, like cerebrospinal fluid (CSF), meninges and eyes. eyes. Several studies have shown promising results and favorable long-term toxicity profiles with this combination. However, the relatively rarity of this tumor precludes rapid completion of large-scale phase III trial and, therefore, our reliance on the results of well-designed phase II trials is critical. Therefore, we evaluate the efficacy and toxicity of thiotepa, bulsulfan, and cyclophosphamide as a conditioning for autologous stem cell transplantation in patients with PCNSL and SCNSL.

ELIGIBILITY:
Inclusion Criteria:

* ∙Patients with histologically confirmed primary central nervous system lymphoma or secondary CNS lymphoma defined as either synchronous CNS involvement of sys- temic NHL or as a site of recurrence in a patient s with a history of systemic NHL

  * Patients who achieved remission after first line chemotherapy and/or WBRT, or who experience relapse of PCNSL/SCNLS.
  * Patients who have not previously received therapy with high high-dose chemotherapy and stem cell transplantatitransplantation.
  * The performance st atus of the patients should be 2 or less by ECOG performance scale.
  * Patients should not have major illness or organ failure incompatible with autologous stem cell transplantation.
* Patients must have adequate hepatic function (serum bilirubin less than 2.0mg/dl, AST and ALT less than three times the upper normal limit)
* Patients must have adequate renal function ( serum creatinin less than 2.0mg/dl)
* Patients must have adequate cardiac function (ejection fraction 45% on echo- cardiogram)
* Patients must have adequate bone marrow function (ANC 1,000/mm 3 and platelet count 75,000/mm 3 ∙ All patients are fully informed about the nature and purpose of this study and informed consent should be given before the start of treatment. All patients should fully understand the right or trial abandon without any disadvantage.

Exclusion Criteria:

* Concurrent history of neoplasm other than CNS lymphoma with life expectancy less than 3 months.
* History of clinically significant cardiac dysfunction (ex. CHF, symptomatic CAD, uncontrolled arrhythmia) or MI within 12 months.
* psychiatric disorders or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible
* significant infection or uncontrolled bleeding
* enrollment of other clinical trials within 4 weeks prior to treatment
* any preexisting medical condition of sufficient severity to prevent full compliance with study
* patient being not willing to or unable to obey study protocol.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 1-year PFS
  PFS was calculated from the date of transplantation to the date of disease progression or death from any cause. Patients who were alive without relapse or progression were censored at the time of last contact.

SECONDARY OUTCOMES:
Overall survival (OS) | through study completion, an average of 1 year
  OS was calculated from the date of transplantation to death from any cause.
Relapse rate | through study completion, an average of 1 year
Non-relapse mortality (NRM) | through study completion, an average of 1 year
  NRM was defined as any death without evidence of relapse.
Toxicity profile | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
not determined